CLINICAL TRIAL: NCT03611062
Title: A Pilot Study on Virtual Reality-based Rehabilitation for Children With Traumatic Brain Injuries
Brief Title: VR-based EF Rehabilitation for Pediatric TBI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Lowell (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Jiabin Shen, PhD, Principal Investigator, University of Massachusetts, Lowell
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: IRB18-00472; 1K99HD093814-01A1 (NIH)
Record Dates: First submitted 2018-06-15; First posted 2018-08-02 (Actual); Results first posted 2021-09-14 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-08

CONDITIONS: Traumatic Brain Injury
Keywords: children; executive function; virtual reality; traumatic brain injury
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR Executive Functions Training (Experimental): Participants will receive training of executive functions in a virtual reality environment.
  Interventions: Behavioral: VR Executive Functions Training
- Control (Placebo Comparator): Participants will play a virtual reality game using the same hardware and similar environments, but without the training of executive functions.
  Interventions: Behavioral: VR Placebo Game

INTERVENTIONS:
Behavioral: VR Executive Functions Training — The Windows 10-based VICT program invites children to rescue an animated character named "Lubdub" from a castle. The program consists of three challenging and child-friendly tasks that correspond to the three core EFs.
  Arms: VR Executive Functions Training
Behavioral: VR Placebo Game — In this game, children in the control group will use the VR hand controller to cast different types of spells (bees, bouncy balls, sparkler spells) to objects in the virtual world. Objects in the VR world will all react differently to a spell being cast so as to provide children a relaxing and EF-free gaming experience.
  Arms: Control

SUMMARY:
Childhood traumatic brain injury (TBI) poses significant impairment in children's executive functions (EFs) for moderate to severe injuries, yet interventions specifically designed for children's EF rehabilitation post-TBI and rigorous clinical trials to establish the safety and efficacy of such interventions remain unavailable. In this study, the investigators will conduct a small-scale pilot randomized clinical trial to evaluate the safety and preliminary efficacy of a novel virtual reality (VR)-based training program for EF rehabilitation for mild complicated to severe childhood TBI. Knowledge from this research will provide empirical evidence for a larger-scale RCT after the conclusion of this pilot study, with the aim to improve the long-term health and quality of life in children with TBI, as well as promote efficiency and effectiveness of future psychological rehabilitation for children with TBI.

DETAILED DESCRIPTION:
Traumatic brain injury (TBI) is a leading cause of acquired disability in U.S. children, with an estimated 700,000 cases every year, presenting in 75% of children with trauma and accounting for 70% of deaths from childhood trauma. Childhood TBIs often result in significant impairment in cognitive functions, particularly in core executive functions (EFs) due to the vulnerability of the frontal lobes, especially after a moderate to severe TBI. Core EF is composed of three skills: inhibitory control, working memory, and cognitive flexibility, whose impairment is associated with impaired daily EF skills, increased attention problems, and lower quality-of-life (QoL). The CDC reported to Congress in 2015 that post-TBI cognitive rehabilitation was the No. 1 unmet health care need for children with TBI. However, evidence-based EF rehabilitation programs are lacking. Although research has shown that a combination of diverse cognitive interventions may improve children's EF, clinically adapting and implementing such interventions in the rehabilitation setting is hampered by limited affordability, accessibility, adherence, and generalizability. Virtual reality (VR) offers an exciting alternative strategy for EF rehabilitation of childhood TBI for three reasons. First, VR has the flexibility to offer various EF training activities in a virtual environment within a restricted physical space. Second, VR can be delivered via Internet/mobile platforms, allowing children to participate in post-discharge training at home as needed. Third, unlike traditional computerized training programs, VR can provide immersive experiences in three dimensions. This may increase adherence to training and foster greater transfer of learned EF skills to untrained tasks in everyday life. Thus far, rigorous randomized clinical trials (RCTs) have not been conducted to establish the safety and efficacy of VR-based EF rehabilitation for childhood TBI.

The overall goal of this pilot project is to assess the feasibility, safety, and preliminary efficacy of a novel VR-based interactive cognitive training (VICT) program for EF rehabilitation in children ages 7-17 years with complicated mild to severe TBI. The VICT program is an integrative hardware and software VR system that trains the three core EFs within a challenging animated mission. Using a small parallel-group RCT, the study focuses on refining clinically-appropriate VR research paradigms in pediatric rehabilitation settings and obtaining feasibility, safety, and preliminary efficacy data on children's EF improvement. After the conclusion of the present pilot study, the investigators will utilize the knowledge and skills gained from this phase to conduct a full-scale longitudinal parallel-group RCT to formally evaluate the VICT program's efficacy.

Specifically, a small parallel-group RCT will be carried out in this study. The investigators aim to recruit 20-30 children with complicated mild to severe TBI and randomly assign each participant to either an intervention group (VICT) or a control group (comparable VR game without EF training). Preliminary efficacy outcomes will be assessed at pre-, post-intervention, and a follow-up visit up to six months after the post-intervention assessment.

Aim 1. Refine clinically-appropriate paradigms for VR childhood TBI rehabilitation research.

Aim 2. Explore feasibility, safety and preliminary efficacy of the VICT program. The feasibility and safety of the VICT program will be examined through both quantitative measures (adverse events, simulator sickness, and fatigability) and a semi-structured interview with children, families, and clinicians regarding perceived benefits and challenges. Preliminary efficacy data will be obtained on core EF, daily EF, attention problems, and health-related QoL for both groups. These data will then be used in a conservative way to estimate the effect size of this novel intervention and calculate the required sample size for future RCTs.

ELIGIBILITY:
Inclusion Criteria:

1. diagnosed with TBI
2. between 7 to 17 years old (inclusive)
3. lowest post-resuscitation Glasgow Coma Scale (GCS)=13-15 combined with trauma-related abnormalities on neuroimaging or a depressed skull fracture (complicated mild TBI, CDC/NIH definition), GCS=9-12 (moderate TBI, CDC/NIH definition), and GCS=3-8 (severe TBI, CDC/NIH definition)
4. fluent in English-based communication
5. currently score <28 on the Agitated Behavior Scale (ABS), indicating mild to no agitation.

Exclusion Criteria:

1. severe physical/visual/cognitive comorbidities secondary to TBI that prevent proper utilization of a VR-based game and valid administration of the study measures
2. premorbid neurological disorder or neurodevelopmental issues prior to injury that prevent proper utilization of a VR-based game and valid administration of the study measures
3. patients who are restricted from using electronic gaming devices.

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 27 (Actual)
Dates: Start 2018-08-15 (Actual); Primary Completion 2020-08-12 (Actual); Study Completion 2020-08-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shen J, Lundine JP, Koterba C, Udaipuria S, Busch T, Rausch J, Yeates KO, Crawfis R, Xiang H, Taylor HG. VR-based cognitive rehabilitation for children with traumatic brain injuries: Feasibility and safety. Rehabil Psychol. 2022 Nov;67(4):474-483. doi: 10.1037/rep0000458. Epub 2022 Jul 21. PMID 35862105

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | VR Executive Functions Training | Control
Started | 14 | 13
Completed | 13 | 12
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | VR Executive Functions Training | Control | Total
Number analyzed (Participants) | 13 | 12 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.77 (3.09) | 11.75 (3.17) | 12.80 (3.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 8 | 8 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 13 | 11 | 24
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 11 | 9 | 20
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Level of Simulator Sickness [Feasibility and Safety]
Description: Measured by the Simulator Sickness Questionnaire. Total scores range from 0 to 26, with 0 representing a better outcome of less sickness.
Time Frame: Post-Intervention, up to 30 minutes after intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | VR Executive Functions Training | Control
Number analyzed (Participants) | 13 | 12
score on a scale | 0.16 (0.19) | 0.03 (0.04)

2. Primary Outcome: Level of Physical Fatigability [Feasibility and Safety]
Description: Measured by the Borg Rating of Perceived Exertion Scale. Total score ranges from 6 to 20, with 6 being a lower amount of exertion.
Time Frame: Post-Intervention, up to 30 minutes after intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | VR Executive Functions Training | Control
Number analyzed (Participants) | 13 | 12
score on a scale | 6.25 (0.50) | 11.50 (2.12)

3. Primary Outcome: Perceived Virtual Reality Experience [Feasibility]
Description: Measured by asking participants to respond to the following question: How much did you like the VR games you just played? Measured on a scale 1-5, with higher values indicating greater enjoyment
Time Frame: Post-Intervention, up to 30 minutes after intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | VR Executive Functions Training | Control
Number analyzed (Participants) | 13 | 12
units on a scale | 3.75 (0.96) | 4 (0)

ADVERSE EVENTS:
Time Frame: During the course of the study participation (up to 30 minutes after study completion)
Arm/Group | VR Executive Functions Training | Control
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/12
Other Adverse Events (participants affected / at risk) | 1/13 | 1/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VR Executive Functions Training (N=13) | Control (N=12)
Blurry vision / eye strain (Eye disorders) | 0 (0) | 1 (1) — reported blurry vision and eye strain after playing part of the virtual reality games. The participant has been seen eye doctors before participating in the study. It was unclear if her pre-condition is related to the reported adverse event.
Headache (General disorders) | 1 (1) | 0 (0) — reported headache after playing part of the virtual reality games.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-04-08): https://cdn.clinicaltrials.gov/large-docs/62/NCT03611062/Prot_SAP_000.pdf
  • Informed Consent Form (2019-04-17): https://cdn.clinicaltrials.gov/large-docs/62/NCT03611062/ICF_001.pdf